CLINICAL TRIAL: NCT05836155
Title: Evidence Based Probiotic Therapy of Proton Pump Inhibitor Induced Gastrointestinal Discomfort and Oralization of the Gut Microbiome: An Open-label Pilot Single-arm Trial
Brief Title: Evidence Based Probiotic Therapy of Proton Pump Inhibitor Induced Dysbiosis
Acronym: EBP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: CBmed Ges.m.b.H. (Other)
Responsible Party: Principal Investigator, Vanessa Stadlbauer-Koellner, MD, Assoc. Prof. PD Dr, Medical University of Graz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 35-175 ex 22/23
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Dysbiosis
MeSH Terms: conditions — Dysbiosis | interventions — Methods

STUDY DESIGN:
Intervention Model Description: unblinded longitudinal study will be performed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The study product contains Bifidobacterium animalis W53, Lactobacillus acidophilus W55, Lactobacillus casei W56, Lactobacillus plantarum W1, Lactobacillus plantarum W21, Lactobacillus rhamnosus W71, and Pediococcus acidilactici W143.
  Interventions: Dietary Supplement: Intervention

INTERVENTIONS:
Dietary Supplement: Intervention — multispecies probiotic

SUMMARY:
In this study the investigators aim to test whether an evidence based probiotic is able to revert proton pump inhibitor induced dysbiosis of the gut microbiome.

DETAILED DESCRIPTION:
With the emergence of high throughput sequencing techniques, researchers obtained the necessary tools to launch in-depth investigations into the structure and function of the intestinal microbiome. For the first time, it was possible to describe the influence of genetics, environment, nutrition and diseases on the microbiome and identify major determinants. One of the most prominent influencing factors on the composition of the microbiome is the use of proton pump inhibitors (PPI), in the general population as well as in chronic diseases, such as liver cirrhosis.

Proton pump inhibitors are used to treat gastric acid related diseases. They drastically reduce the secretion of gastric acid and thereby increase the gastric pH. The reduction of gastric acid production, however, allows acid-sensitive food-borne and oral bacteria to pass the stomach unharmed and colonize the more distal parts of the intestine. In addition, PPI use creates less favorable conditions for typical gut commensals and reduces the microbial diversity in the intestine. These alterations in the microbiome can be linked to PPI side effects, such as gastrointestinal symptoms (e.g., abdominal discomfort, bloating, constipation or diarrhea) and an increased risk for enteral infections. In patients with liver cirrhosis, PPI-induced changes in the microbiome, namely Streptococcus salivarius and Veillonella parvula - two oral bacteria, are linked to intestinal inflammation and gut permeability and predict a higher risk of complications and a higher three-year liver related mortality. These are considerable risks that need to be weighed against the benefits of the therapy. Reduction of PPI use to cases with a clear indication is one important measure to reduce potential harm of the treatment. However, many patients require long-term treatment, e.g. for gastroesophageal reflux disease or to prevent gastrointestinal bleeding when drugs with a high risk of bleeding are used (such as thrombocyte aggregation inhibitors and oral anticoagulation). Therefore, strategies to reduce oralization and thereby symptoms and negative consequences of PPI are necessary.

One possibility to change the composition of the gut microbiome is the use of probiotic bacteria. Probiotics are live microorganisms that have been demonstrated to alter the gut microbiome and exhibit positive effects on numerous gastrointestinal complaints, strengthen the gut barrier and reduce inflammation parameters. The investigators previously showed in a pilot study that a multispecies probiotic was able to improve gut permeability biomarkers in patients with long-term PPI therapy as well as gastrointestinal symptoms. However, this product was not able to efficiently reverse oralization. Therefore, the investigators conducted a series of experiments, including direct and indirect pathogen inhibition tests to identify probiotic strains that are capable of inhibiting the growth of Streptococcus salivarius and Veillonella parvula in vitro to design an evidence based probiotic mixture. The investigators screened 43 QPS (Qualified presumption of safety, granted by the European Food Safety Authority) certified probiotic strains and identified 5 strains as potential therapeutic agents to prevent/treat PPI induced oralization (unpublished data).

ELIGIBILITY:
Inclusion Criteria:

* Age >18;
* Signed Informed Consent;
* PPI intake for at least 3 months;
* Willing to accept use of all encoded data, including publication, and the confidential use and storage of all data for at least 15 years; Exclusion criteria
* Diagnosed with a gastrointestinal infection within 4 weeks prior to screening; Severe gastrointestinal disorders (e.g. inflammatory bowel diseases)
* Received any of the following products/medication prior to screening: systemic antibiotics, prokinetics, prebiotic supplements, probiotic supplements within 4 weeks prior to screening;
* Concomitant diseases or other circumstances that suggest that the patients are not eligible for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Changes in overall symptom score | 3 months
  Gastrointestinal quality of life index (GIQLI)

SECONDARY OUTCOMES:
Other dimension of gastrointestinal quality of life | 3 months
  Gastrointestinal quality of life index (GIQLI)
Composition of the faecal metabolome | 3 months
  NMR metabolomics
Zonulin | 3 months
  measurement of faecal zonulin
Calprotectin | 3 months
  measurement of faecal calprotectin
Diaminooxidase | 3 months
  measurement of serum diaminooxidase
lipopolysaccharide binding protein | 3 months
  measurement of serumlipopolysaccharide binding protein
soluble CD14 | 3 months
  measurement of serum soluble CD14
Veillonella parvula | 3 months
  measurement of stool Veillonella parvula gene abundance
Streptococcus salivarius | 3 months
  measurement of stool Streptococcus salivarius gene abundance

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
Microbiome data will be shared in a public repository, other data will depend on results and IPR discussions between partners
Supporting Information: Study Protocol, SAP
Time Frame: Microbiome data will be shared in a public repository when the paper will be submitted, other data will depend on results and IPR discussions between partners